CLINICAL TRIAL: NCT03114124
Title: Microfidelity (MIFI) Ablation Technology Versus Standard Ablation Catheter for Atrioventricular Nodal Ablation A Comparative Pilot Study of Time to Success
Brief Title: Microfidelity (MIFI) Ablation Technology Versus Standard Ablation Catheter for Atrioventricular Nodal Ablation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ir-iis02
Record Dates: First submitted 2017-03-21; First posted 2017-04-14 (Actual); Results first posted 2021-09-01 (Actual); Last update posted 2021-09-22 (Actual); Status verified 2021-08

CONDITIONS: Atrial Fibrillation
Keywords: ablation; atrioventricular node; microfidelity
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Intervention Model Description: Standard ablation catheter vs MIFI catheter
Who Masked: Investigator
Masking Description: Variable block sizes will be used to improve the blinding of the clinical team. This information will then be used to design a fully-powered randomized study to compare these two arms. Patients will be randomly assigned to study arms. The project biostatistician and team will generate a set of envelopes which contain the random assignments for each patient. Once a patient has consented to participate, the next envelope will be opened for that patient and the catheter assignment will be revealed. This will maintain the blinding of the clinical team.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Bipolar Ablation Catheter (Active Comparator): Subjects will be randomized by random computer programming to receive standard ablation catheter for their procedure.
  Interventions: Device: Standard Ablation Catheter
- MIFI Ablation Catheter (Experimental): Subjects will be randomized by random computer programming to receive an ablation with MIFI technology. MIFI Catheter contains tightly spaced multielectrode pattern
  Interventions: Device: MIFI Catheter

INTERVENTIONS:
Device: MIFI Catheter — Multielectrode Catheter: standard ablation catheter that has the ability to record low and high frequency signals with high fidelity
  Arms: MIFI Ablation Catheter
Device: Standard Ablation Catheter — Standard of care for patients with certain cardiac arrhythmias.
  Arms: Bipolar Ablation Catheter

SUMMARY:
The aim of our study is to investigate the comparative efficacy of high fidelity multi electrode ablation catheters vs the standard bipolar configuration in success of AV nodal ablation This study will provide insights on the use of new technology where application may increase efficacy, promote patient and physician safety and decrease costs.

DETAILED DESCRIPTION:
Introduction In some elderly patients with atrial fibrillation (AF), especially in combination with heart failure, a rate control strategy may be preferred. When pharmacological therapy is ineffective or not tolerated, it is reasonable to perform atrioventricular (AV) node ablation with ventricular pacing as a class IIA indication per current guidelines.

Usually, the procedure is simple and straightforward and complete heart block can be achieved without any difficulty. However, this "simple" procedure can sometimes prove to be a most difficult case. The most common reason for failure to achieve complete heart block is the inability to localize the compact AV node using the His signal with standard intracardiac electrograms. As these patients come to the laboratory in AF, the His signal may be obscured by AF waves. In some patients with a deeper intramyocardial location of the His bundle and compact AV node it becomes necessary to produce deeper ablation lesions using an irrigated catheter to achieve block.

In patients with AF, the target of ablation for the "ablate and pace" approach is the compact AV node, located at the apex of the triangle of Koch. Ideally, ablation is performed at the most proximal penetrating part of the His bundle in order to maintain a proximal automatic junctional rhythm and avoid pacemaker dependence.

Para Hisian pacing is most commonly used to reveal the presence of a septal accessory pathway.

The His bundle is a deep insulated structure and it is difficult to capture it at usual energy outputs. Using a high- output pacing (usually 20 mA at 2 msec) it is possible to directly capture the deeply situated His bundle, which is confirmed by a narrower QRS complex on the paced electrograms. Thus, high-output pacing can be utilized to map the His bundle area in difficult situations.

By applying this electrophysiologic principle of differential tissue capture to help identify the location of the compact AV node, which is in close proximity to the His bundle. Ventricular pacing was performed initially at high output to capture both the basal right ventricular myocardium and the His bundle and the output was gradually lowered to lose His bundle capture. The QRS duration is relatively narrow with high output pacing and increases when the pacing output is lowered, representing ventricular myocardial capture alone. Finally, loss of ventricular capture is seen with further reduction of pacing output. This maneuver has been shown to aid in determining the proximity of the ablation catheter to compact AV node as was validated by successful ablation at this site. Parahisian pacing in conjunction with av nodal ablation has recently been described in the literature.

A novel catheter with three mini electrodes within the ablation tip (IntellaTip MiFi, Boston Scientific, Boston, MA) may enhance the available data for such a signal dependent technique. In this catheter, bipolar signals can be recorded between the three 0.8-mm-wide electrodes that are arranged radially 1.3 mm from the end of the catheter alongside the standard distal and proximal bipolar recordings. Animal studies have already demonstrated that the mini electrodes in this novel catheter are more accurate in identifying conducting gaps in linear ablations than conventional electrode recordings.

Study Aims:

The aim of our study is to investigate the comparative efficacy of high fidelity multi electrode ablation catheters vs the standard bipolar configuration in success of AV nodal ablation This study will provide insights on the use of new technology where application may increase efficacy, promote patient and physician safety and decrease costs.

Primary and secondary objectives Primary endpoints

1. Acute success of ablation identified by a junctional rhythm or complete heart block
2. Time from application of radiofrequency energy to acute success

Secondary endpoints include

1. Procedure time
2. Radiation time
3. Frequency of ablation application
4. Duration of ablation application

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a diagnosis of persistent or permanent atrial fibrillation documented on electrocardiography
2. Patients must meet American College of Cardiology and Heart Rhythm Society "ACC/HRS" guidelines for atrioventricular nodal ablation procedure
3. Patients must be available for at least 1 month post procedure
4. Patients must be greater than or equal to 18 years old.

Exclusion Criteria:

1. Patients who do not meet ACC/HRS indications for av nodal ablation

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-05-23 (Actual); Primary Completion 2019-09-26 (Actual); Study Completion 2019-11-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John N Catanzaro, MD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: There was no wash out or run-in event. The significant portion of the research was the AV nodal ablation
Period: Overall Study
Arm/Group | Bipolar Ablation Catheter | MIFI Ablation Catheter
Started | 15 | 15
Completed | 15 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bipolar Ablation Catheter | MIFI Ablation Catheter | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 2 | 4
  >=65 years | 13 | 13 | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 75.8 (11.09) | 72.46 (10.4) | 74.13 (10.73)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 4 | 10
  Male | 9 | 11 | 20
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 15 | 15 | 30

OUTCOME MEASURES:

1. Primary Outcome: The Time Differences Between the 2 Arms for Acute Success of Ablation Identified by a Junctional Rhythm or Complete Heart Block
Description: Identified by a junctional rhythm or complete heart block. Time zero is when the ablation procedure begins and the successful outcomes are either complete heart block or junctional rhythm.
Time Frame: 60 seconds
Population: Randomized
Measure: Median (Inter-Quartile Range); unit: seconds
Arm/Group | Bipolar Ablation Catheter | MIFI Ablation Catheter
Number analyzed (Participants) | 15 | 15
seconds | 5 [3 to 16] | 4 [1 to 5]

2. Secondary Outcome: Time From Application of Radio-frequency Energy to Acute Success
Description: The target will be where the HIS electrogram amplitude is greatest and where the QRS complex from pacing is narrowest.
Time Frame: up to 3000 seconds
Population: Randomized
Measure: Median (Inter-Quartile Range); unit: seconds
Arm/Group | Bipolar Ablation Catheter | MIFI Ablation Catheter
Number analyzed (Participants) | 15 | 15
seconds | 615 [277 to 2778] | 525 [110 to 1371]

ADVERSE EVENTS:
Time Frame: 2 weeks
Arm/Group | Bipolar Ablation Catheter | MIFI Ablation Catheter
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-01-25): https://cdn.clinicaltrials.gov/large-docs/24/NCT03114124/Prot_SAP_002.pdf